CLINICAL TRIAL: NCT06150989
Title: A Biobehavioral Approach to Understand the Multilevel Determinants of Cardiovascular Health in Black Women
Brief Title: Black Women's Life Experience On Cardiovascular Health Via Ongoing Monitoring
Acronym: BLOOM
Status: Recruiting | Type: Observational
Sponsor: The University of Texas at Arlington (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Yue Liao, Assistant Professor, The University of Texas at Arlington
Other Study IDs: 2023-0344
Record Dates: First submitted 2023-10-20; First posted 2023-11-30 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Heart Disease Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Group: Black women enrolled in this study will complete a series of lab-based assessments that evaluate their vascular health, followed by a 10-day free-living monitoring period with mobile and wearable devices.
  Interventions: Behavioral: Observational Group

INTERVENTIONS:
Behavioral: Observational Group — All participants will go through a series of lab-based assessments to evaluate their vascular health. These assessments include: heart rhythm/rate, blood pressure, large blood vessel flow, central aortic blood pressure and pulse wave velocity, brain blood flow, carbon dioxide concentration, flow mediated dilation/blood vessel responsiveness, breathing rate, and cerebral vasomotor reactivity. In addition, venous blood sample will be taken to identify biomarkers that are associated with elevating blood pressure and decreasing blood flow.
  The 10-day monitoring period includes a wrist-worn activity tracker and a blood pressure monitor bracelet; a smartphone app that will prompt surveys up to 6 times a day to assess behaviors, social/physical context, mood/stress, and experience of racial discrimination/microaggression. Participants will also collect saliva samples on three consecutive days during the 10-day monitoring period.

SUMMARY:
This pilot study uses a state-of-the-science combination of remote behavioral monitoring, real-time experience sampling, in-lab physiological assessments, and extraction of neighborhood-level characteristics to (1) Examine the impact of daily experience (i.e., racial discrimination, affective states, stress) on health behaviors (i.e., physical activity, sedentary behavior, sleep) at the intrapersonal level among Black women; (2) Test the association between daily behaviors and impairments in biomarkers associated with vascular function/health (i.e., augmented systemic inflammation and oxidative stress, impaired peripheral/cerebral vascular function, increased large artery stiffness), as well as the impact of daily experience on the relationship between behaviors and vascular function; and (3) Explore the influence of neighborhood-level characteristics (i.e., social environment factors: i.e., neighborhood income and poverty, racial composition; and built environment context, such as park density and walkability) on daily experience and health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* born and identified as female;
* between 18-49 years old;
* self-identify as Black or African American;
* not currently pregnant;
* ownership of a smartphone with Internet access;
* able to speak and read English

Exclusion Criteria:

* diagnosed hypertension, cardiovascular, respiratory, metabolic, and/or neurological disorders;
* functional limitations or health issues that preclude physical activity;
* currently taking medications for thyroid function or psychological conditions such as depression, anxiety, and mood disorders;
* current use of oral or inhalant corticosteroids for asthma;
* have regularly smoked within the last 2 years.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The target population for this study is non-pregnant Black women between the ages of 18 to 49.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Macrovascular function | Day 1
  Macrovascular function will be assessed as brachial artery vasodilation following a period of suprasystolic cuff occlusion. Microvascular function will be assessed as the % change in blood velocity from baseline following cuff release.
Arterial Stiffness | Day 1
  An appropriately sized blood pressure cuff will be placed on the upper arm and central (aortic) and peripheral (arm) blood pressure will be assessed using the non-invasive SphygmoCor Xcel device. This device provides measurement of augmentation index (in percentage), which is an indicator of arterial stiffness.
Blood Flow Measurements (Large Blood Vessels) | Day 1
  A Doppler ultrasound probe will be used to measure blood flow in the upper arm, leg, and/or neck (e.g., brachial artery, femoral artery, and carotid artery, respectively).
Blood Flow Measurements (Cerebral Blood Vessels) | Day 1
  Cerebral blood flow will be indexed from the velocity of blood flowing through the middle cerebral artery. This will be accomplished using transcranial Doppler ultrasound.

SECONDARY OUTCOMES:
Physical activity | Day 2 to Day 11
  Daily physical activity level will be assessed via a wrist-worn accelerometer.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level study data will be deposited to the ICPSR, an AHA-approved data repository, for sharing behavioral health and social science research data. Codebooks (or data dictionaries) and other study documentation will be made available as PDFs on the ICPSR website.

REFERENCES:
- [Derived] Liao Y, Brothers RM, Brown KK, Lee RE. A biobehavioral observational study to understand the multilevel determinants of cardiovascular health in Black women: the BLOOM Study protocol. BMC Womens Health. 2024 Jul 5;24(1):391. doi: 10.1186/s12905-024-03182-0. PMID 38970037